CLINICAL TRIAL: NCT00502645
Title: SINGLE-CENTER,OPEN,NON-CONTROLLED FEASIBILITY STUDY ON THE PERFORMANCE OF THE CS-1 DECISION SUPPORT SYSTEM WITH INCORPORATED SOFTWARE-ALGORITHM eMPC USED FOR BLOOD GLUCOSE CONTROL OVER 72 HOURS IN CRITICALLY ILL PATIENTS AT THE INTENSIVE CARE UNIT
Brief Title: Clinical Risk Assesment of CS-1 Decision Support System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM10_CS-1
Record Dates: First submitted 2007-07-15; First posted 2007-07-17 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-07

CONDITIONS: Hyperglycemia; Critically Ill Patients
Keywords: algorithm; cs-1 decision support system; insulin; hyperglycemia; tight glycemic control; intensive care; adults
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CS-1 DECISION SUPPORT SYSTEM

SUMMARY:
This is a single-center, open, non-controlled clinical investigation in 10 patients at the Medical University Graz including a treatment visit (V1)and a follow up visit(V2). In the treatment visit (V1) after admittance to the ICU arterial blood glucose values will be monitored and either the software-algorithm eMPC will be used to adjust the infusion rate of intravenously administered human soluble insulin to normalise arterial blood glucose. The purpose of the present study is to investigate the performance of the already developed and tested algorithm in combination with a newly developed bed-side, touch screen user interface (CS-1 decision support system) in patients at the medical ICU for a period of 72 hours. Follow up information(V2) will be acquired at hospital discharge or at the latest one week after visit 1.

DETAILED DESCRIPTION:
Before the beginning of any trial related activities, the relatives of each patient will be asked if the patient has ever mentioned in the past, that he/she does not want do participate in any kind of clinical study. If this was said by the patient in the past or if there are any signs which make it likely that the patient would not participate, he/she will be excluded from the trial. After testing of the inclusion and exclusion criteria, screening information will be obtained a the beginning of the trial. A screening number will be assigned to the patient in ascending order. The following data will be recorded in the case record form (CRF): Check for inclusion/exclusion criteria,demographic data, medical (including diabetes) history and relevant medication, body weight and heightand laboratory analyses from routine laboratory assessment. Patients fulfilling all the inclusion criteria and none of the exclusion criteria will be included into the trial and a subject number will be assigned in ascending order. Routine intensive care will be provided from department of internal medicine. Trial related activities will not interfere with regular patient care. Blood samples will be retrieved from an arterial line, available for routine diagnostic and monitoring procedures in all patients. At time 0, a blood glucose measurement will be taken, manually entered into the CS-1 decision support system and both a insulin infusion rate and the time to next glucose reading will be suggested by the computer-based system. Based on the suggestion of the system, an insulin infusion pump as routinely used in the ICU will be manually set to this suggested insulin infusion rate by specially trained ICU staff but only if the staff feels safe with this suggestion. Intravenous infusion of human soluble insulin will then be started. For safety reasons: In case that the suggested measurement interval of the decision support system exceeds a 90 minute interval, interim glucose measurements will be taken. All measurements will be documented in the CRF. Only in case that the blood glucose values are below 40 mg/dl the additional interim-glucose value will also be put into the CS-1 system. However, the nursing staff can at any time decide to take an additionlal blood glucose measurement and/or neglect the decision as suggested by the system.

The target range for blood glucose levels will be 80-110 mg/dl [4.4 - 6.1 mmol/l]. The current blood glucose level and insulin infusion rate will continuously be documented by the CS-1 decision support system and supervised by the investigator. Glucose values will be provided to the system by manual entry. In case of hypoglycaemia, intravenous insulin infusion will be stopped and glucose will be administered via intravenous bolus.

The treatment visit, including all trial related activities as described above, will last for 72 hours. Adverse events and relevant medication will be continuously monitored and documented The Acute Physiology and Chronic Health Evaluation Score (Apache II) will be documented for each patient at the beginning of the trial. There is no physical connection between the algorithm suggesting the insulin infusion rate and the insulin infusion pump such as that the algorithm would be capable to independently steer the insulin infusion. There is also no physical connection between the glucose measurement device and the algorithm such as that the algorihthm would be able to independently get a glucose measurement. For safety reasons, both the glucose measurement and the insulin infusion rate are parameters that need to be manually entered by a specially trained nurse. For glucose measurement, a certified device for ICU application is being used (Accuchek® Inform; Roche Diagnostics), for intravenous insulin infusion, a certified insulin infusion pump (Perfusor® Space, BBraun Melsungen) as it is used under routine conditions in the ICU is being used. Follow up information will be acquired at hospital discharge or at the latest one week after visit 1. .

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years of age
* Stay in the ICU expected to be > 72 h
* Blood glucose > 110 mg/dl or patient on insulin treatment

Exclusion Criteria:

* Patients with hyperglycaemic crisis/ketoacidosis due to insulin deficiency.
* Known or suspected allergy to insulin
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient (i.e., liver failure, other fatal organ failures)
* Patients participating in another study
* Moribund patients likely to die within 24 hours
* Patients after organ transplantation within the last three months
* Patients under high dose cortisol treatment (cortisol > 1000 mg/day or equivalent dosis of hydrocortisol)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percentage of time within predefined glucose target range 80-110mg/dL | Start: Start of treatment ; End: Last glucose measurement under treatment

SECONDARY OUTCOMES:
Hypoglycemias (<40mg/dl =2,2mM); Blood sampling frequency as adviced by device; Malfunctions of device Relevant-medication, nutrition; Insulin Infusion Rate; Blood glucose values; Handling/ usability of device; | Start: Start of treatment, End: Last glucose measurement under treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Austria

REFERENCES:
- [Background] Plank J, Blaha J, Cordingley J, Wilinska ME, Chassin LJ, Morgan C, Squire S, Haluzik M, Kremen J, Svacina S, Toller W, Plasnik A, Ellmerer M, Hovorka R, Pieber TR. Multicentric, randomized, controlled trial to evaluate blood glucose control by the model predictive control algorithm versus routine glucose management protocols in intensive care unit patients. Diabetes Care. 2006 Feb;29(2):271-6. doi: 10.2337/diacare.29.02.06.dc05-1689. PMID 16443872